CLINICAL TRIAL: NCT05630755
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Clinical Study to Evaluate a Switch to Doravirine/Islatravir (DOR/ISL 100 mg/0.25 mg) Once-Daily in Participants With HIV-1 Who Are Virologically Suppressed on Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF)
Brief Title: A Switch to Doravirine/Islatravir (DOR/ISL) in Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Who Are Virologically Suppressed on Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) (MK-8591A-052)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8591A-052; MK-8591A-052 (Other: MSD); 2022-502079-49-00 (Registry Identifier: EU CT); jRCT2051230003 (Registry Identifier: jRCT); U1111-1283-0949 (Registry Identifier: UTN)
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — doravirine; islatravir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DOR/ISL and Placebo to BIC/FTC/TAF (Experimental): Participants will receive DOR/ISL 100 mg/0.25 mg and Placebo to BIC/FTC/TAF once daily (QD) orally from day 1 to week 144. After week 144, eligible participants may continue on DOR/ISL and continue study treatment until week 240 or to when DOR/ISL becomes commercially accessible (whichever comes first).
  Interventions: Drug: DOR/ISL; Drug: Placebo to BIC/FTC/TAF
- BIC/FTC/TAF and Placebo to DOR/ISL (Active Comparator): Participants will receive BIC/FTC/TAF 50 mg/200 mg/25 mg and Placebo to DOR/ISL once daily (QD) orally from day 1 to week 144. After week 144, eligible participants may switch to DOR/ISL and continue study treatment until week 240 or to when DOR/ISL becomes commercially accessible (whichever comes first).
  Interventions: Drug: BIC/FTC/TAF; Drug: Placebo to DOR/ISL

INTERVENTIONS:
Drug: DOR/ISL — DOR/ISL 100 mg/0.25 mg oral tablets once daily
  Other Names: MK-8591A; Doravirine/Islatravir
  Arms: DOR/ISL and Placebo to BIC/FTC/TAF
Drug: BIC/FTC/TAF — BIC/FTC/TAF 50 mg/200 mg/25 mg oral tablets once daily
  Other Names: Bictegravir/Emtricitabine/Tenofovir Alafenamide
  Arms: BIC/FTC/TAF and Placebo to DOR/ISL
Drug: Placebo to BIC/FTC/TAF — 0 mg oral tablets once daily
  Arms: DOR/ISL and Placebo to BIC/FTC/TAF
Drug: Placebo to DOR/ISL — 0 mg oral tablets once daily
  Arms: BIC/FTC/TAF and Placebo to DOR/ISL

SUMMARY:
The primary objectives of this study are to evaluate the antiretroviral activity of a switch to Doravirine/Islatravir (DOR/ISL) compared with continued Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) at Week 48; and to evaluate the safety and tolerability of a switch to DOR/ISL compared with continued BIC/FTC/TAF, through Week 48. The primary hypotheses are that (1) DOR/ISL is non-inferior to continued BIC/FTC/TAF, as assessed by the percentage of participants with HIV-1 ribonucleic acid (RNA) ≥50 copies/mL at Week 48, with a margin of 4 percentage points used to define non-inferiority; and (2) DOR/ISL is superior to BIC/FTC/TAF, as assessed by the percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 48.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Is HIV-1 positive with plasma HIV-1 RNA <50 copies/mL
* Has been receiving BIC/FTC/TAF therapy with documented viral suppression (HIV-1 RNA <50 copies/mL) for ≥3 consecutive months prior to providing documented informed consent and has no history of prior virologic treatment failure on any past or current regimen
* Female is not a participant of childbearing potential (POCBP); or if a participant of childbearing potential, not pregnant or breastfeeding, and is willing to use an acceptable contraceptive method or abstain from heterosexual intercourse for study duration

Exclusion Criteria:

* Has HIV-2 infection
* Has a diagnosis of an active acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within 30 days prior to screening
* Has active hepatitis B virus (HBV) infection
* Has chronic hepatitis C virus (HCV) infection with laboratory values consistent with cirrhosis
* Has a history of malignancy ≤5 years prior to providing documented informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or cutaneous Kaposi's sarcoma
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or strong and moderate cytochrome P450 3A (CYP3A) inducers
* Has a documented or known virologic resistance to DOR
* Has taken long-acting HIV therapy at any time (e.g., cabotegravir, lenacapavir)
* Is currently participating in or has participated in a clinical study and received (or is receiving) an investigational compound or device from 45 days prior to Day 1 through the study treatment period except those currently enrolled in the comparator arm of an ongoing DOR/ISL study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2028-08-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (49):
- United States (24):
  - Pueblo Family Physicians ( Site 1425), Phoenix, Arizona
  - Pacific Oaks Medical Group ( Site 1400), Beverly Hills, California
  - Ruane Clinical Research Group, Inc ( Site 1414), Los Angeles, California
  - Mills Clinical Research ( Site 1433), Los Angeles, California
  - Whitman-Walker Institute ( Site 1431), Washington D.C., District of Columbia
  - Therafirst Medical Center ( Site 1402), Fort Lauderdale, Florida
  - Midway Immunology and Research Center ( Site 1401), Ft. Pierce, Florida
  - AHF The Kinder Medical Group ( Site 1426), Miami, Florida
  - Orlando Immunology Center ( Site 1407), Orlando, Florida
  - Triple O Research Institute, P.A ( Site 1417), West Palm Beach, Florida
  - Infectious Disease Specialists of Atlanta ( Site 1403), Decatur, Georgia
  - Mercer University, Department of Internal Medicine ( Site 1411), Macon, Georgia
  - AccessHealth MA ( Site 1419), Boston, Massachusetts
  - Be Well Medical Center ( Site 1408), Berkley, Michigan
  - KC CARE Health Center-Clinical Trials ( Site 1422), Kansas City, Missouri
  - Las Vegas Research Center ( Site 1436), Las Vegas, Nevada
  - Regional Center for Infectious Disease Research ( Site 1435), Greensboro, North Carolina
  - Central Texas Clinical Research ( Site 1413), Austin, Texas
  - St Hope Foundation ( Site 1410), Bellaire, Texas
  - Prism Health North Texas, Oak Cliff Health Center ( Site 1409), Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A ( Site 1404), Dallas, Texas
  - Texas Centers for Infectious Disease Associates ( Site 1406), Fort Worth, Texas
  - The Crofoot Research Center ( Site 1424), Houston, Texas
  - DCOL Center for Clinical Research ( Site 1415), Longview, Texas
- Australia (5):
  - Holdsworth House Medical Practice ( Site 6200), Darlinghurst, New South Wales
  - St Vincent's Hospital-IBAC ( Site 6203), Sydney, New South Wales
  - Holdsworth House Medical Practice - Brisbane ( Site 6201), Brisbane, Queensland
  - Royal Brisbane and Women's Hospital-Infectious Diseases Research ( Site 6204), Brisbane, Queensland
  - Prahran Market Clinic ( Site 6202), Melbourne, Victoria
- Chile (4):
  - Clinica Universidad Catolica del Maule ( Site 2204), Talca, Maule Region
  - Clínica Universidad de Los Andes ( Site 2206), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile-Inmunologia Alergia y VIH ( Site 2200), Santiago, Region M. de Santiago
  - Hospital hernan henriquez aravena de temuco-Unidad de Investigación Clínica ( Site 2205), Temuco, Región de la Araucanía
- Israel (4):
  - Rambam Health Care Campus-Institute of Allergy, Clinical Immunology, ( Site 4801), Haifa
  - Hadassah Medical Center-Infecious Disease ( Site 4802), Jerusalem
  - Sheba Medical Center-HIV unit ( Site 4803), Ramat Gan
  - Sourasky Medical Center ( Site 4804), Tel Aviv
- Japan (3):
  - National Hospital Organization Nagoya Medical Center ( Site 6603), Nagoya, Aichi-ken
  - Center Hospital of the National Center for Global Health and Medicine ( Site 6601), Shinjyuku-ku, Tokyo
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research ( Site 66, Osaka
- United Kingdom (9):
  - Southmead Hospital ( Site 5805), Bristol, Bristol, City of
  - Queen Elizabeth Hospital Birmingham ( Site 5809), Birmingham, England
  - Royal Liverpool University Hospital ( Site 5812), Liverpool, England
  - Royal London Hospital ( Site 5800), London, England
  - Royal Free Hospital ( Site 5801), London, England
  - Guy's & St Thomas' NHS Foundation Trust ( Site 5808), London, London, City of
  - The Mortimer Market Centre for Sexual Health and HIV Research ( Site 5810), London, London, City of
  - University Hospital of Wales ( Site 5803), Cardiff, Wales
  - Royal Berkshire Hospital ( Site 5813), Reading

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Colson AE, Mills AM, Ramgopal MN, Bettacchi C, Osiyemi OO, Hinestrosa F, Crofoot G, Katner HP, Gatanaga H, Johnson M, Diamond TL, Barninger E, Eves K, Su FH, Xu Y, Klopfer SO, Stamm LM, Fox MC, Lahoulou R. Switch to fixed-dose doravirine (100 mg) and islatravir (0.25 mg) once daily in virologically suppressed adults with HIV-1 on bictegravir, emtricitabine, and tenofovir alafenamide: 48-week results of a phase 3, multicentre, randomised, controlled, double-blind, non-inferiority trial. Lancet. 2026 Feb 7;407(10528):611-621. doi: 10.1016/S0140-6736(25)01948-8. PMID 41654375
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26114&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- DOR/ISL and Placebo to BIC/FTC/TAF: Participants will receive doravirine/islatravir (DOR/ISL) 100 mg/0.25 mg and Placebo to bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) once daily (QD) orally from day 1 to week 144. After week 144, eligible participants may continue on DOR/ISL and continue study treatment until week 240 or to when DOR/ISL becomes commercially accessible (whichever comes first).
Period: Overall Study
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Started | 343 | 171
Treated | 342 | 171
Completed | 10 | 6
Not Completed | 333 | 165
Not completed — Lost to Follow-up | 7 | 0
Not completed — Randomized by Mistake Without Study Treatment | 1 | 0
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Participant moved away from trial site | 0 | 1
Not completed — Status not Recorded | 316 | 161

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL | Total
Number analyzed (Participants) | 343 | 171 | 514
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (12.9) | 47.6 (13.1) | 47.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 36 | 110
  Male | 269 | 135 | 404
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 44 | 117
  Not Hispanic or Latino | 262 | 125 | 387
  Unknown or Not Reported | 8 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 20 | 10 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 112 | 47 | 159
  White | 206 | 106 | 312
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) ≥50 Copies/mL at Week 48
Description: HIV-1 RNA levels in blood samples taken at each visit were measured with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: The analysis population includes all randomized participants who received ≥1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Number analyzed (Participants) | 342 | 171
Percentage of Participants | 1.5 | 0.6
Statistical Analysis 1: Comparison: DOR/ISL and Placebo to BIC/FTC/TAF vs BIC/FTC/TAF and Placebo to DOR/ISL; Test type: Non-Inferiority — A margin of 4 percentage points is used to define non-inferiority; p = 0.003, Miettinen and Nurminen method; Unstratified Miettinen and Nurminen method was used; Risk Difference (RD) = 0.88, 95% CI 2-sided [-1.86 to 2.90]; The estimated difference was calculated using the unstratified Miettinen and Nurminen method
Statistical Analysis 2: Comparison: DOR/ISL and Placebo to BIC/FTC/TAF vs BIC/FTC/TAF and Placebo to DOR/ISL; Test type: Superiority; p = 0.192, Miettinen and Nurminen method; Unstratified Miettinen and Nurminen method was used; Risk Difference (RD) = 0.88, 95% CI 2-sided [-1.86 to 2.90]; The estimated difference was calculated using the unstratified Miettinen and Nurminen method

2. Primary Outcome: Percentage of Participants Who Experience Adverse Events (AEs) Through Week 48
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE is reported.
Time Frame: Up to Week 48
Population: The analysis population includes all randomized participants who received ≥1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Number analyzed (Participants) | 342 | 171
Percentage of Participants | 74.6 | 71.3

3. Primary Outcome: Percentage of Participants Who Discontinue Study Intervention Due to AEs Through Week 48
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE is reported.
Time Frame: Up to Week 48
Population: The analysis population includes all randomized participants who received ≥1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Number analyzed (Participants) | 342 | 171
Percentage of Participants | 2.9 | 1.8

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 48
Description: HIV-1 RNA levels in blood samples taken at each visit were measured with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <200 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: The analysis population includes all randomized participants who received ≥1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Number analyzed (Participants) | 342 | 171
Percentage of Participants | 91.8 | 94.2

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48
Description: HIV-1 RNA levels in blood samples taken at each visit were measured with a reliable lower limit of quantification of <50 copies/mL. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: The analysis population includes all randomized participants who received ≥1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Number analyzed (Participants) | 342 | 171
Percentage of Participants | 91.5 | 94.2

6. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4-positive (CD4+) T-cell Count at Week 48
Description: Plasma CD4+ T-Cell Count was measured in cells/mm^3 for baseline and 48 weeks. Baseline measurements were defined as the Day 1 value of each participant. The change from baseline to Week 48 and corresponding 2-sided 95% confidence intervals were calculated based on cLDA models adjusted by treatment group, time, and the interaction of time-by-treatment group.
Time Frame: Baseline at Day 1 and Week 48
Population: The analysis population includes all randomized participants who received ≥1 dose of study intervention and who had baseline data for CD4+ T-cell count.
Measure: Mean (95% Confidence Interval); unit: Cells/mm^3
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Number analyzed (Participants) | 315 | 161
Cells/mm^3 | 30.40 [10.98 to 49.83] | 28.19 [-4.46 to 60.83]

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent, Resistance-associated Substitutions at Week 48
Description: Participants with clinically significant confirmed viremia [2 consecutive occurences 4 weeks (+-1 week) apart of HIV-1 RNA ≥200 copies/mL at any time during the study] or who discontinue study intervention for another reason with HIV-1 RNA ≥200 copies/mL at the time of discontinuation met the criteria for post-baseline resistance testing. Per protocol, participants with HIV-1 RNA ≥400 copies/mL or any participant for whom available genotypic or phenotypic data show evidence of resistance, irrespective of viral load were included in the resistance analysis subset. Plasma samples were collected for genotypic and phenotypic HIV-1 viral drug resistance testing and used to assess resistance-associated substitutions and virus susceptibility to study intervention. The percentage of participants in the resistance analysis subset with treatment-emergent resistance-associated substitutions to the study intervention is presented.
Time Frame: Up to Week 48
Population: Per protocol, participants with HIV-1 RNA ≥400 copies/mL or any participant for whom available genotypic or phenotypic data show evidence of resistance, irrespective of viral load were included in the resistance analysis subset. Participants without available assay results were not included.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
Number analyzed (Participants) | 1 | 0
Percentage of Participants | 0 |

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥50 Copies/mL at Week 96
Description: Percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 96 will be reported.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2029-08

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 96
Description: Percentage of participants with HIV-1 RNA <200 copies/mL at Week 96 will be reported.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2029-08

10. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 96
Description: Percentage of participants with HIV-1 RNA <50 copies/mL at Week 96 will be reported.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2029-08

11. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 96
Description: Mean change from baseline at Day 1 in CD4+ T-cell count at Week 96 will be reported.
Time Frame: Baseline at Day 1 and Week 96
Reporting Status: Not Posted, anticipated posting 2029-08

12. Secondary Outcome: Number of Participants With Viral Drug Resistance Mutations at Week 96
Description: Number of participants with evidence of viral drug resistance-associated substitutions at Week 96 will be reported.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2029-08

13. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥50 Copies/mL at Week 144
Description: Percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 144 will be reported.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2029-08

14. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 144
Description: Percentage of participants with HIV-1 RNA <200 copies/mL at Week 144 will be reported.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2029-08

15. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 144
Description: Percentage of participants with HIV-1 RNA <50 copies/mL at Week 144 will be reported.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2029-08

16. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 144
Description: Mean change from baseline at Day 1 in CD4+ T-cell count at Week 144 will be reported.
Time Frame: Baseline at Day 1 and Week 144
Reporting Status: Not Posted, anticipated posting 2029-08

17. Secondary Outcome: Number of Participants With Viral Drug Resistance Mutations at Week 144
Description: Number of participants with evidence of viral drug resistance-associated substitutions at Week 144 will be reported.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2029-08

18. Secondary Outcome: Percentage of Participants Who Experience AEs Through Week 144
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Week 144
Reporting Status: Not Posted, anticipated posting 2029-08

19. Secondary Outcome: Percentage of Participants Who Discontinue Study Intervention Due to AEs Through Week 144
Description: as for outcome 18
Time Frame: Up to Week 144
Reporting Status: Not Posted, anticipated posting 2029-08

ADVERSE EVENTS:
Time Frame: Up to 84 weeks
Description: All-cause mortality (ACM): all randomized participants; AEs: all randomized participants who received at least one dose of study treatment.
Arm/Group | DOR/ISL and Placebo to BIC/FTC/TAF | BIC/FTC/TAF and Placebo to DOR/ISL
All-Cause Mortality (participants affected / at risk) | 0/343 | 0/171
Serious Adverse Events (participants affected / at risk) | 15/342 | 11/171
Other Adverse Events (participants affected / at risk) | 94/342 | 52/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/ISL and Placebo to BIC/FTC/TAF (N=342) | BIC/FTC/TAF and Placebo to DOR/ISL (N=171)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/ISL and Placebo to BIC/FTC/TAF (N=342) | BIC/FTC/TAF and Placebo to DOR/ISL (N=171)
Diarrhoea (Gastrointestinal disorders) | 20 (21) | 6 (6)
Fatigue (General disorders) | 13 (13) | 12 (12)
COVID-19 (Infections and infestations) | 21 (22) | 9 (9)
Influenza (Infections and infestations) | 9 (9) | 9 (10)
Nasopharyngitis (Infections and infestations) | 21 (25) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (26) | 8 (8)
Dizziness (Nervous system disorders) | 11 (11) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT05630755/Prot_SAP_000.pdf